CLINICAL TRIAL: NCT05098106
Title: PlaIaR-Trial: Platelets in Inflammation and Resolution.
Acronym: PLAIAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Study Chair and Principal Investigator: Univ.-Prof. Dr. Alexander Zarbock (Unknown); Principal Investigator: Dr. Andreas Margraf (Unknown)
Responsible Party: Sponsor
Other Study IDs: 12-Anit-20
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: ARDS; Platelet Abnormality
MeSH Terms: conditions — Blood Platelet Disorders | interventions — Bronchoscopy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage fluid, blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pneumonia patients with ARDS: Patients in the perioperative/intensive care setting with pneumonia-induced ARDS requiring bronchoscopy.
  Interventions: Diagnostic Test: Bronchoscopy, blood sampling; testing.
- Ventilated patients without ARDS: Patients without ARDS on mechanical ventilation.
  Interventions: Diagnostic Test: Bronchoscopy, blood sampling; testing.

INTERVENTIONS:
Diagnostic Test: Bronchoscopy, blood sampling; testing. — BAL and blood samples are measured by hematology analyzer, flow cytometry, western blot, RNAseq analysis and multiplex.

SUMMARY:
Detection and determination of platelets in bronchoalveolar lavage fluid and blood in ARDS and non-ARDS-patients. Correlation with phenotype and inflammation parameters in blood and outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* Routine bronchoscopy
* Patient in perioperative setting
* Age >=18 years
* Consent

Exclusion Criteria:

* Active or recent (in past 7 days) bleeding in upper airways
* Recent traumatic injury of the lung associated with (micro-)hemorrhage
* Blood aspiration
* Pregnancy
* Age<18 years
* Acute kidney injury / Chronic kidney failure / Dialysis
* Transplantation
* HIV
* Hematologic diseases
* Immunosuppression
* Anti-Platelet-Therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Perioperative patients
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Detectability and changes in platelets in BAL and blood | 5-7 days
Organ failure, survival. | 1 Year
Systemic platelet and leukocyte numbers | 5-7 days
Systemic platelet and leukocyte phenotypes. | 5-7 days
Systemic cytokine profiles. | 5-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zarbock, Univ.-Prof. Dr., Study Chair — University Hospital Muenster; Andreas Margraf, Dr., Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, Germany

IPD SHARING:
Plan to Share IPD: Undecided